CLINICAL TRIAL: NCT06717204
Title: Vericiguat for Ventricular Remodeling in Patients With Heart Failure With Reduced Ejection Fraction After Myocardial Infarction
Brief Title: Vericiguat for Heart Failure With Reduced Ejection Fraction After Myocardial Infarction
Acronym: HFrEF
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Jinan Central Hospital (Other); Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Pan-Pan Hao, Professor, Qilu Hospital of Shandong University
Other Study IDs: Vericiguat for HFrEF
Record Dates: First submitted 2024-12-01; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: HFrEF - Heart Failure With Reduced Ejection Fraction; Myocardial Infarction (MI)
Keywords: HFrEF; Myocardial Infarction; Vericiguat
MeSH Terms: conditions — Myocardial Infarction | interventions — vericiguat; Prescription Drugs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vericiguat and conventional treatment: Vericiguat in addition to conventional treatment
  Interventions: Drug: Vericiguat Oral Tablet [Verquvo]; Drug: Prescription Drugs
- Conventional treatment only: Conventional treatment only
  Interventions: Drug: Prescription Drugs

INTERVENTIONS:
Drug: Vericiguat Oral Tablet [Verquvo] — Vericiguat in addition to conventional treatment
  Other Names: Conventional treatment
  Groups: Vericiguat and conventional treatment
Drug: Prescription Drugs — Conventional treatment only
  Other Names: Conventional treatment without vericiguat

SUMMARY:
The effects of vericiguat on cardiac remodeling in patients with chronic stable heart failure after myocardial infarction have not been reported. This project aims to clarify the efficacy and safety of vericiguat in patients with chronic heart failure after myocardial infarction. Patients with chronic stable heart failure with reduced ejection fraction after myocardial infarction in the electronic medical records of Qilu Hospital of Shandong University will be selected and divided into two groups: the treatment group received vericiguat in addition to conventional treatment and the control group received conventional treatment only. After 12-month treatment, the effects of vericiguat on cardiac remodeling and function and cardiovascular adverse events will be evaluated. The results are helpful to provide a new treatment strategy for chronic heart failure after myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

1. The history of acute myocardial infarction exceeds 3 months;
2. Symptoms and signs of heart failure have been stable for more than one month;
3. 18 years old or more;
4. NYHA cardiac function classified as grade II~IV;
5. LVEF≤40%；
6. NT-proBNP≥450pg/ml；
7. All subjects or their guardians must sign the subject consent before entering the trial.

Exclusion Criteria:

1. Patients with the following diseases: nonischemic cardiomyopathy; valvular heart disease; congenital heart disease; obstruction of left ventricular outflow tract; severe decompensated heart failure; active myocarditis or pericardial disease; end-stage liver and kidney diseases; malignant tumor;
2. Mechanical complications of myocardial infarction;
3. Unable to obtain primary outcome data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic heart failure with reduced ejection fraction after myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
LVEDVI=LVEDV/BSA | From baseline to the end of 12-month treatment
  Changes of left ventricular end-diastolic volume index (LVEDVI) compared with baseline after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Panpan Hao, MD, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (3):
- China (3):
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - The First Affiliated Hospital of Shandong First Medical University/Shandong Province Qianfoshan Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Undecided
Institutional policy and patient privacy.